CLINICAL TRIAL: NCT06251661
Title: Cognitive Multi-sensory Rehabilitation on Upper Limb Functions and Fatigue in Different Grades of Spasticity in Stroke Patients
Brief Title: Cognitive Multi-sensory Rehabilitation on Upper Limb Function and Fatigue in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gehad Mohamed Mohamdeen Ali Mohamed, Lecturer Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMR stroke
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Ischemic
Keywords: CMR; Stroke; upper limb function; fatigue
MeSH Terms: conditions — Stroke; Ischemia; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (GA) (Active Comparator): 20 Egyptian ischemic stroke patients receive 12 sessions of CMR and traditional physical therapy each session lasts for 40 minutes of CMR and 30 minutes of traditional physical therapy.
  Interventions: Other: Cognitive multi-sensory Rehabilition; Other: selected traditional physical therapy program.
- Group 2 (GB) (Sham Comparator): 20 Egyptian ischemic stroke patients receive 12 sessions of traditional physical therapy each session lasts for 30 minutes.
  Interventions: Other: selected traditional physical therapy program.

INTERVENTIONS:
Other: Cognitive multi-sensory Rehabilition — Kinetic awareness: Initially, only one joint will be moved at a time. Then the therapist will reposition the joint and ask the participants to report their perception of the joint position. Initially, the participants will distinguish between just two positions. If they reliably answer correctly, increase up to five points and integrate speed and dexterity in functional movements. Participants will be asked to relax and feel the movement during this training. Discrimination exercise: The therapist places a part of the participant's limb, the fingertip, on an external object (a block) and the participant will be asked to actively move his or her limb over the object and try to sense the shape of the object. If the participants differentiate between the two objects, then increase the number of objects (up to five). Functional training: The patient reaches toward many objects functionally (cup, ball, cane) from different angles, holds them, and relocates them again.
  Arms: Group 1 (GA)
Other: selected traditional physical therapy program. — The selected physical therapy program session will be occupational therapy training for the hand, strengthening exercises for the weak upper limb stretching exercises for short upper limb muscles, balance exercise, and gait training.

SUMMARY:
This interventional study aims to investigate the therapeutic efficacy of Cognitive multi-sensory rehabilitation (CMR) on upper limb function and fatigue in chronic stroke patients. The main question is:

• Does cognitive multi-sensory rehabilitation significantly affect upper limb function and fatigue in stroke patients? Participants will be assigned into two groups. They will receive 12 sessions of study group CMR and traditional physical therapy and control group traditional physical Therapy rehabilitation. CMR 40 minutes immediately followed by 20 minutes of selected physical therapy program, three sessions per week for four weeks.

DETAILED DESCRIPTION:
About 70% of people with stroke are unable to use their affected hand efficiently in activities of daily living. Further, post-stroke fatigue affects up to 92% of post-stroke patients. Post-stroke fatigue is a multifaceted motor and cognitive process, in which the patient experiences tiredness and lack of energy that develops during physical or mental activity which may persist for years. Post-stroke fatigue impacts the mental/physical functions of the patient through decreased energy, and thus, is a significant barrier to recovery.

Preliminary evidence indicates sensory rehabilitation may enhance motor recovery in people with stroke. Cognitive Multisensory Rehabilitation (CMR) is a therapist-guided sensorimotor rehabilitation approach, that targets the patients' ability to solve sensory discrimination exercises, where the patient compares the sensations felt by the hand to the shapes observed with the eyes. Cognitive processes are encouraged by asking the patient to determine the limb movement or its position, how the movement was felt in the body, how the limb moved in relation to other parts of the body, and to spatial parameters in the environment. Because CMR integrates cognitive processes with sensory and motor tasks, it may be a novel method to address post-stroke fatigue, and it may increase connectivity in sensory and motor areas of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 65 years.
* 6-18 months after ischemic stroke
* living in the community (i.e., not in a long-term care home).
* medically stable.
* normal score in the Montreal Cognitive Assessment (MoCA: 25 to 30, maximum score = 30).
* Spasticity of upper limb muscles ranged from (grade 1:2) according to the Modified Ashworth scale.

Exclusion Criteria:

* severe spasticity (Modified Ashworth Scale score of 4)
* any medical condition that hinders full participation,
* another neurological diagnosis beyond stroke including cognitive impairment, or
* upper extremity pain > 4/10 on the Numeric Pain Rating Scale (maximum 10/10).

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be applied to ischemic stroke. This type of stroke is more common in males than females because most smokers are males. As known, smoking is the major cause of ischemic stroke due to atherosclerotic changes in cerebral blood vessels.
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for upper extremity (FMT-UE). | from baseline to four weeks after the beginning of intervention
  Changes in upper limb function.
Serum levels of Brain-Derived Neurotrophic Factor (BDNF) | from baseline to four weeks after the beginning of intervention
  Changes in serum levels of neural plasticity factors
Changes in hand grip strength | from baseline to four weeks after the beginning of intervention
  Hand grip strength was measured by an electronic hand dynamometer device.
Fatigue Assessment Scale (FAS) | from baseline to four weeks after the beginning of intervention
  determine the degree of self-reported fatigue in daily living activities.
  Each item of the FAS is answered using a fi ve-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Items 4 and 10 are reverse-scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.

SECONDARY OUTCOMES:
Box and Blocks Test (BBT) | from baseline to four weeks after beginning of the intervention.
  Changes in gross hand function intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nahed Salem, professor, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Giza Governorate, Egypt